CLINICAL TRIAL: NCT05309590
Title: Prospective Pilot Study Evaluating the Efficacy of Low-Dose Topical Steroids in Maintaining Histologic Remission of Eosinophilic Esophagitis in Children
Brief Title: Efficacy of Low-Dose Topical Steroids in Maintaining Remission of Eosinophilic Esophagitis in Children
Status: Active, not recruiting | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Joshua Wechsler, Principal Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2014-15753
Record Dates: First submitted 2022-01-24; First posted 2022-04-04 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dose Reduction: All patients recruited to the study will have reduced their swallowed steroid medication from twice to once daily as part of the standard-of-care.
  Interventions: Drug: Dose

INTERVENTIONS:
Drug: Dose — The outcomes of reducing to half of the topical steroid (i.e. fluticasone [Flovent] and Swallowed viscous budesonide [Pulmicort]) will be observed with regards to whether the patients continue to be in histologic remission. These patients will have already achieved remission on a full dose of the steroid.

SUMMARY:
This study evaluates the decrease in steroid dosing for patients who have achieved remission on a full dose of steroids. Once a patient is in remission they will be enrolled in this study if they choose to decrease the steroid dosing.

DETAILED DESCRIPTION:
As the disease usually recurs once steroids are discontinued, and there is concern for complications of untreated disease, continuation of steroids is indefinite after induction of remission. The short-term safety of topical steroids has been well established; however, long-term safety has not been studied in EoE. Concerns for long-term complications of chronic steroid therapy include effects on bone density and stature as has been suggested by literature in patients with asthma treated with inhaled corticosteroids chronically.4, 5 It remains unclear whether symptom and histologic remission, once achieved, can be maintained with a lower, to be defined, dosage of topical steroids.6 This is critical to prevent the major complications associated with uncontrolled eosinophilic inflammation: fibrotic remodeling (scarring) of the esophagus and eventual stricture (narrowing of the esophagus).7-11

Several studies have demonstrated that remission with induction (approximately 3 months of therapy) dose topical steroids resulted in resolution of inflammation and concurrent reversal of sub-epithelial early-stage fibrosis.12-18 It has not, however, been established whether fibrosis recurs when patients are maintained on induction doses long-term or whether lower "maintenance" dosing is sufficient. Studies are therefore needed to demonstrate whether fibrosis can be prevented from recurring long-term, ideally at a lower maintenance dose to minimize potential complications of therapy. Therapeutic strategies that achieve continuous and sustained remission with resolution of eosinophilic inflammation will prevent chronic symptoms along with remodeling, fibrosis and eventual esophageal stricture.

The rationale for utilizing lower dose topical steroids for maintaining clinical and histologic remission in children is the potential to lower the steroid-related side effects including contracting oral and/or esophageal fungal infections (a yeast infection which causes white patches in the mouth and throat), loss of bone density, suppression of adrenal-cortical axis (turns off the body's usual production of cortisol, which helps the body maintain a balance and respond to stress), and failure to achieve linear growth (height) potential. There are no studies that have properly quantified the risk of swallowed steroids in EoE, thus the investigators are presuming and postulating a lower cumulative risk of adverse effects from long-term use of the medication with this lower dose than the standard dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with EoE
* Patients less than 21 years of age at enrollment
* Patients who within the past 12 months have demonstrated histologic remission (<15 eos/hpf as assessed by upper esophagogastroduodenoscopy (EGD) with biopsy ) to the standard induction dose of topical steroids and have remained on this treatment:

  * Topical steroid treatment includes only those with previously published results: Swallowed topical fluticasone (i.e. Flovent®), and Swallowed viscous budesonide (i.e. Pulmicort Respules®) mixed with Honey or Splenda®
* Patients who are interested in lowering their dose of topical steroids.

Exclusion Criteria:

* Patients with EoE who have not demonstrated histologic remission (<15 eos/hpf) to topical steroids.
* Patients who are unable or unwilling to take topical steroids.
* Patients who have changed the vehicle or carrier (e.g. Splenda®or honey ) used to mix with the actual steroid drug, after demonstrating histologic remission.

Ages: 1 Year to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: By design, this study involves the participation of children. It is not anticipated that any other special groups be enrolled in a proportion other than that representative of the US population. Enrollment will not be limited by race or gender.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Low Dose Topical Steroid | At standard of care endoscopies from the date of enrollment; estimated every 6-12 months
  Number of patients who maintain histologic remission of low dose (50% dosing) topical steroids

SECONDARY OUTCOMES:
Visual and histologic assessment of the esophagus | At standard of care endoscopies from the date of enrollment; estimated every 6-12 months
  assess the change in visual findings on steroid or half dose steroid and whether patients were able to maintain visual and histologic remission when on low dose (50% dosing) topical steroids

CONTACTS AND LOCATIONS:
Overall Officials: Joshua B Wechsler, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Childjren's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schoepfer AM, Safroneeva E, Bussmann C, Kuchen T, Portmann S, Simon HU, Straumann A. Delay in diagnosis of eosinophilic esophagitis increases risk for stricture formation in a time-dependent manner. Gastroenterology. 2013 Dec;145(6):1230-6.e1-2. doi: 10.1053/j.gastro.2013.08.015. Epub 2013 Aug 13. PMID 23954315
- [Background] Dellon ES, Kim HP, Sperry SL, Rybnicek DA, Woosley JT, Shaheen NJ. A phenotypic analysis shows that eosinophilic esophagitis is a progressive fibrostenotic disease. Gastrointest Endosc. 2014 Apr;79(4):577-85.e4. doi: 10.1016/j.gie.2013.10.027. Epub 2013 Nov 23. PMID 24275329
- [Background] Papadopoulou A, Koletzko S, Heuschkel R, Dias JA, Allen KJ, Murch SH, Chong S, Gottrand F, Husby S, Lionetti P, Mearin ML, Ruemmele FM, Schappi MG, Staiano A, Wilschanski M, Vandenplas Y; ESPGHAN Eosinophilic Esophagitis Working Group and the Gastroenterology Committee. Management guidelines of eosinophilic esophagitis in childhood. J Pediatr Gastroenterol Nutr. 2014 Jan;58(1):107-18. doi: 10.1097/MPG.0b013e3182a80be1. PMID 24378521
- [Background] Weldon D. The effects of corticosteroids on bone growth and bone density. Ann Allergy Asthma Immunol. 2009 Jul;103(1):3-11; quiz 11-3, 50. doi: 10.1016/S1081-1206(10)60135-4. PMID 19663120
- [Background] de Vreede I, Haarman EG, Sprikkelman AB, van Aalderen WM. From knemometry to final adult height: inhaled corticosteroids and their effect on growth in childhood. Paediatr Respir Rev. 2013 Jun;14(2):107-11; quiz 111, 137-8. doi: 10.1016/j.prrv.2012.05.001. Epub 2012 Jun 9. PMID 23718991
- [Background] Liacouras CA, Furuta GT, Hirano I, Atkins D, Attwood SE, Bonis PA, Burks AW, Chehade M, Collins MH, Dellon ES, Dohil R, Falk GW, Gonsalves N, Gupta SK, Katzka DA, Lucendo AJ, Markowitz JE, Noel RJ, Odze RD, Putnam PE, Richter JE, Romero Y, Ruchelli E, Sampson HA, Schoepfer A, Shaheen NJ, Sicherer SH, Spechler S, Spergel JM, Straumann A, Wershil BK, Rothenberg ME, Aceves SS. Eosinophilic esophagitis: updated consensus recommendations for children and adults. J Allergy Clin Immunol. 2011 Jul;128(1):3-20.e6; quiz 21-2. doi: 10.1016/j.jaci.2011.02.040. Epub 2011 Apr 7. PMID 21477849
- [Background] Straumann A, Bussmann C, Zuber M, Vannini S, Simon HU, Schoepfer A. Eosinophilic esophagitis: analysis of food impaction and perforation in 251 adolescent and adult patients. Clin Gastroenterol Hepatol. 2008 May;6(5):598-600. doi: 10.1016/j.cgh.2008.02.003. Epub 2008 Apr 14. PMID 18407800
- [Background] Fox VL, Nurko S, Teitelbaum JE, Badizadegan K, Furuta GT. High-resolution EUS in children with eosinophilic "allergic" esophagitis. Gastrointest Endosc. 2003 Jan;57(1):30-6. doi: 10.1067/mge.2003.33. PMID 12518127
- [Background] Kwiatek MA, Hirano I, Kahrilas PJ, Rothe J, Luger D, Pandolfino JE. Mechanical properties of the esophagus in eosinophilic esophagitis. Gastroenterology. 2011 Jan;140(1):82-90. doi: 10.1053/j.gastro.2010.09.037. Epub 2010 Sep 19. PMID 20858491
- [Background] Chehade M, Sampson HA, Morotti RA, Magid MS. Esophageal subepithelial fibrosis in children with eosinophilic esophagitis. J Pediatr Gastroenterol Nutr. 2007 Sep;45(3):319-28. doi: 10.1097/MPG.0b013e31806ab384. PMID 17873744
- [Background] Aceves SS, Newbury RO, Dohil R, Bastian JF, Broide DH. Esophageal remodeling in pediatric eosinophilic esophagitis. J Allergy Clin Immunol. 2007 Jan;119(1):206-12. doi: 10.1016/j.jaci.2006.10.016. PMID 17208603
- [Background] Wagener JS, Wojtczak HA. Inhaled steroids in children: risks versus rewards. J Pediatr. 1998 Mar;132(3 Pt 1):381-3. doi: 10.1016/s0022-3476(98)70003-4. No abstract available. PMID 9544884
- [Background] Aceves SS, Bastian JF, Newbury RO, Dohil R. Oral viscous budesonide: a potential new therapy for eosinophilic esophagitis in children. Am J Gastroenterol. 2007 Oct;102(10):2271-9; quiz 2280. doi: 10.1111/j.1572-0241.2007.01379.x. Epub 2007 Jun 20. PMID 17581266
- [Background] Straumann A, Degen L, Felder S, et al. Budesonide As Induction Treatment for Active Eosinophilic Esophagitis In Adolescents and Adults: A Randomized, Double-Blind, Placebo-Controlled Study (Bee-I Trial). Gastroenterology 2008;134:A-104.
- [Background] Dohil R, Newbury R, Fox L, Bastian J, Aceves S. Oral viscous budesonide is effective in children with eosinophilic esophagitis in a randomized, placebo-controlled trial. Gastroenterology. 2010 Aug;139(2):418-29. doi: 10.1053/j.gastro.2010.05.001. Epub 2010 May 7. PMID 20457157
- [Background] Straumann A, Conus S, Degen L, Felder S, Kummer M, Engel H, Bussmann C, Beglinger C, Schoepfer A, Simon HU. Budesonide is effective in adolescent and adult patients with active eosinophilic esophagitis. Gastroenterology. 2010 Nov;139(5):1526-37, 1537.e1. doi: 10.1053/j.gastro.2010.07.048. Epub 2010 Aug 1. PMID 20682320
- [Background] Aceves SS, Newbury RO, Chen D, Mueller J, Dohil R, Hoffman H, Bastian JF, Broide DH. Resolution of remodeling in eosinophilic esophagitis correlates with epithelial response to topical corticosteroids. Allergy. 2010 Jan;65(1):109-16. doi: 10.1111/j.1398-9995.2009.02142.x. Epub 2009 Oct 1. PMID 19796194
- [Background] Straumann A, Conus S, Degen L, Frei C, Bussmann C, Beglinger C, Schoepfer A, Simon HU. Long-term budesonide maintenance treatment is partially effective for patients with eosinophilic esophagitis. Clin Gastroenterol Hepatol. 2011 May;9(5):400-9.e1. doi: 10.1016/j.cgh.2011.01.017. Epub 2011 Jan 28. PMID 21277394
- [Background] Pappa H, Thayu M, Sylvester F, Leonard M, Zemel B, Gordon C. Skeletal health of children and adolescents with inflammatory bowel disease. J Pediatr Gastroenterol Nutr. 2011 Jul;53(1):11-25. doi: 10.1097/MPG.0b013e31821988a3. PMID 21694532
- [Background] Miheller P, Lorinczy K, Lakatos PL. Clinical relevance of changes in bone metabolism in inflammatory bowel disease. World J Gastroenterol. 2010 Nov 28;16(44):5536-42. doi: 10.3748/wjg.v16.i44.5536. PMID 21105186
- [Background] Schmidt S, Mellstrom D, Norjavaara E, Sundh V, Saalman R. Longitudinal assessment of bone mineral density in children and adolescents with inflammatory bowel disease. J Pediatr Gastroenterol Nutr. 2012 Nov;55(5):511-8. doi: 10.1097/MPG.0b013e31825817a0. PMID 22688562